CLINICAL TRIAL: NCT01057056
Title: The Role of Mind Body Therapy in Geriatric Rehabilitation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Yaffa Lerman, Director ,Geriatrics Division. Dr Shahar Lev-ari, Acting manager; complementary medicine unit, Tel-Aviv Sourasky Medical Center
Purpose: Supportive Care
Other Study IDs: TASMC-09-YL-0488-CTIL; 0488-09-TLV (Other: tel-aviv medical center)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-01

CONDITIONS: Elderly; Treatment
Keywords: patients in a sub-acute geriatric rehabilitation department

ARMS (1):
- control group (No Intervention): control group - receiving standard treatment
  Interventions: Other: mind-body intervention

INTERVENTIONS:
Other: mind-body intervention — multi-disciplinary mind-body intervention including: breathing techniques, guided imagery, meditation, touch therapy

SUMMARY:
Background: The main goal of geriatric rehabilitation reconditioning following an acute illness is rapid restoration of normal activity. Key elements are pain control, restoration of bowel functions, sleep, appetite and general well-being, along side the physical activity.

Objective: To assess the effect of mind-body intervention as an adjunct to medical and physical rehabilitation in geriatric patients.

Design: Prospective study Setting: University affiliated large city general hospital

ELIGIBILITY:
Inclusion Criteria:

* suitable candidates had to be aged 18 years or older
* treated in the Geriatric Rehabilitation Department in the Tel Aviv Sourasky Medical Center (TASMC) and
* were willing and able to complete the study protocol.

Exclusion Criteria:

* severe unstable chronic illness (e.g., congestive heart failure, chronic renal failure, cancer).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2010-01

PRIMARY OUTCOMES:
Well-being: Short Form-36 (SF-36), Geriatric Depression Scale (GDS)